CLINICAL TRIAL: NCT01216826
Title: Phase II Study of Everolimus in Children and Adolescents With Refractory or Relapsed Osteosarcoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sidnei Epelman (Other)
Responsible Party: Sponsor-Investigator, Sidnei Epelman, Director of Pediatric Oncology Department, Hospital Santa Marcelina
Organization: Hospital Santa Marcelina (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001CBR07T
Record Dates: First submitted 2010-10-04; First posted 2010-10-07 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Refractory or Relapsed Osteosarcoma
MeSH Terms: conditions — Osteosarcoma | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Everolimus (Experimental)
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — Everolimus will be administered every day, initial dose 5 mg/m²/dia, in 28 days cycles. Maximum dosis: 10 mg/day. The cycles will be repeated till progression disease or untolerable toxicity.
  Other Names: Afinitor, RAD.

SUMMARY:
The purpose of this study is to determine the Everolimus aim response in children and adolescents with refractory or relapsed osteosarcoma.

The aim response is defined as complete or partial response (according to RECIST criteria) for at least 4 weeks, or stable disease for at least 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Osteosarcoma histological confirmation.
* No option of known curative treatment, neither approved treatment that increases survival with adequate quality of life.
* Karnofsky scale ≥ 50 for patients over 16 years and Lansky scale ≥ 50 for patients under 16 years.
* Subjects should not have received antineoplastic therapy < 4 weeks before study treatment initiation.
* Adequate hematological function: neutrophil count > 1.500/mm³, platelets > 100.000/mm³ and hemoglobin > 8.0 mg/dL.
* Adequate renal function, as defined below:

Age Maximum serum creatinine (mg/dL) 0 - 29 days 0,4 - 0,7 1 month - 3 years 0,7 4 - 7 years 0,8 8 - 10 years 0,9 11 - 12 years 1,0 13 - 17 years 1,2

≥18 years 1,3

* Adequate hepatic function: total bilirubin ≤ 1.5 x ULN and transaminases ≤ 2.5 x ULN.
* Patient and/or legal responsible must sign ICF.
* Life expectation > 8 weeks.
* Measurable disease, according to RECIST criteria.
* For female patients of childbearing age: Presence of a negative pregnancy test within 7 days prior to day 0.
* The patient agrees to use effective contraception if procreative potential exists. Use of reliable means of contraception (e.g. hormonal contraceptive, patch, vaginal ring, intrauterine device, physical barrier, abstinence) for subjects of reproductive potential (males and females) is required during study treatment and for 3 months following last dose of study drug

Exclusion Criteria:

* History of myocardial infarction, angina or cerebrovascular accident related to atherosclerosis.
* Pulmonary disorder (e.g. FEV1 or DLCO ≤ 70% upper expected).
* Significant hematologic or hepatic abnormality (transaminases levels > 2.5 x ULN or serum bilirubin >1.5 x ULN, hemoglobin < 8 g/dL, platelets < 100.000/ mm3, ANC < 1.500/mm3).
* Has other existing serious medical conditions that could adversely affect the ability of the patient to be treated in accordance with the protocol.
* Any condition, therapy, or medical condition, which, in the opinion of the attending physician could represent a risk for the patient or adversely affect the study objectives.
* If female, is pregnant or lactating.
* Active infection at the moment of recruitment.
* Previous history of organ transplantation.
* Recent surgery < 2 months before entering study.
* Concomitant antineoplastic therapy.
* Patient received more than one rescue treatment, previously.
* Previous treatment with mTor inhibitors (ex: sirolimus, temsirolimus, everolimus).
* Use of investigational drug < 30 days before entering study.
* Non-controlled hyperlipidaemia: serum cholesterol (fasting) > 300 mg/dL or 7,75 mmol/L and triglycerides (fasting) > 2,5 x ULN.
* Non-controlled diabetes mellitus defined as: glycemia (fasting) > 1.5 x ULN.
* Patient with hemorrhagic disorder or using oral anti-vitamin K (except warfarin in low doses).
* Patient with HIV infection.
* Incapable to perform protocol visits.
* Another neoplasia for the last 2 years (except squamous or basocellular skin cancer).
* Hypersensitivity history to rapamycin analogs.
* Chronic treatment with corticoids (except per oral, topical or local treatment) or another immunosuppressor agent.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-03; Primary Completion 2014-06 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Determine the Everolimus aim response in children and adolescents with refractory or relapsed osteosarcoma | Up to 2 years.

SECONDARY OUTCOMES:
Define Everolimus toxicity in this population | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Sidnei Epelman, MD, Principal Investigator — Hospital Santa Marcelina
Locations (1):
- Hospital Santa Marcelina, São Paulo, São Paulo, Brazil